CLINICAL TRIAL: NCT05492760
Title: Evaluation of Recurrence Risk of Atrial Fibrillation After Cryoballoon Ablation： a Retrospective Cohort Study
Brief Title: Evaluation of Recurrence Risk of Atrial Fibrillation After Cryoballoon Ablation
Acronym: era-cryo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, professor, Shanghai 10th People's Hospital
Other Study IDs: era-cryo
Record Dates: First submitted 2022-07-31; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ablation group
  Interventions: Device: cryoballoon ablation

INTERVENTIONS:
Device: cryoballoon ablation — Patients with AF will accept cryoballoon ablation.

SUMMARY:
The recurrence of atrial fibrillation(AF) after pulmonary vein ablation with cryoballoon is conducted by many factors . The previous studies found larger left atrial and longer AF duration are tied to higher risk of AF recurrence. The characters of ablation procedure is also of critical importance to durable clinical success such as temperature features and time-to-isolation (TTI). The aim of our study is to develop an tool of recurrence risk evaluation with both pre-procedure and procedure factors.

ELIGIBILITY:
Inclusion Criteria:

Patients with paroxysmal AF and accept cryoballoon ablation.

Exclusion Criteria:

* left atrium (LA) diameter (anterior-to-posterior)>55mm on transthoracic echocardiography (TTE)
* the presence of thrombus in the LA or left atrial appendage (LAA) on transesophageal echocardiography (TEE)
* uncorrected heart failure (NYHA class III or IV),
* concomitant moderate or severe valvular heart disease or bioprosthetic valve,
* malignancy necessitating chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal AF and accept cryoballoon ablation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
the time to atrial fibrillation recurrent | 1year after the cryoballoon ablation
  the time to atrial fibrillation recurrent

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, doctor, Study Director — Shanghai 10th People's Hospital

IPD SHARING:
Plan to Share IPD: No